CLINICAL TRIAL: NCT00719732
Title: Visual Function After Implantation of Bilateral AcrySof ReSTOR Aspheric +3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Diane Houtman, Alcon Research, Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M07-001; NCT00762203 (obsolete NCT alias)
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Cataract
Keywords: ReSTOR Aspheric +3 IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReSTOR Aspheric +3 (Experimental): Enrolled subjects receive implantation of ReSTOR +3 intraocular lenses (IOLs) for replacement of cataract in the natural lens of the eye. The patients were to be implanted bilaterally (in both eyes).
  Interventions: Device: ReSTOR

INTERVENTIONS:
Device: ReSTOR — Enrolled subjects receive implantation of ReSTOR +3 intraocular lenses (IOLs) for replacement of cataract in the natural lens of the eye. The patients were to be implanted bilaterally (in both eyes).

SUMMARY:
A prospective evaluation of the visual parameters in a series of patients bilaterally implanted with AcrySof ReSTOR +3 Intraocular Lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cataracts

Exclusion Criteria:

* Pre-existing conditions that could skew the results or are contraindications for the ReSTOR intraocular lens;
* <1 diopter astigmatism by keratometry readings.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 18 - 70 years of age, either sex and any race. Diagnosis of cataracts in one or both eyes.
Pre-assignment Details: Subject's eligibility was determined at the preoperative visit. All subjects met inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | ReSTOR Aspheric +3
Started | 218
Completed | 196
Not Completed | 22
Not completed — Lost to Follow-up | 20
Not completed — Unilateral (not bilateral) implantation | 1
Not completed — Illness not associated with device | 1

BASELINE CHARACTERISTICS:
Arm/Group | ReSTOR Aspheric +3
Number analyzed (Participants) | 218
Age Categorical [Number; unit: participants] — Date of birth received for 207 of 218 subjects; therefore, age data not available for 11 subjects.
  participants
    <=18 years | 0
    Between 18 and 65 years | 143
    >=65 years | 64
Gender [Number; unit: participants] — Gender not received for 212 of 218 subjects, therefore, gender missing for 6 subjects.
  participants
    Female | 88
    Male | 124

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Visual Acuity (UCVA)
Description: Uncorrected Visual Acuity (UCVA) measured by means of logMAR at various distances (40 centimeters (cm), 50 cm, 60 cm, 70 cm, and 4 meters (m)). Visual Acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Aspheric +3
Number analyzed (Participants) | 196
logMAR
  UCVA at 40 cm | 0.05 (0.10)
  UCVA at 50 cm | -0.07 (0.15)
  UCVA at 60 cm | 0.15 (0.14)
  UCVA at 70 cm | 0.20 (0.13)
  UCVA at 4 m | -0.01 (0.11)

ADVERSE EVENTS:
Time Frame: Up to 6 months post-operative
Description: Volunteered and solicited adverse events were collected from the time of surgery to the 6 month post-operative visit.
Arm/Group | ReSTOR Aspheric +3
Serious Adverse Events (participants affected / at risk) | 1/196
Other Adverse Events (participants affected / at risk) | 0/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReSTOR Aspheric +3 (N=196)
Chronic inflammation/iritis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Condfidential information will be submitted for publication without Sponsor's prior written agreement.